CLINICAL TRIAL: NCT00173797
Title: Comparison of Psychometric Properties of Three Depression Measures in Patients With Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9361701232; NSC-94-2314-B-002-080
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-07

CONDITIONS: Cerebrovascular Accidents
Keywords: depression; psychometrics
MeSH Terms: conditions — Stroke; Depression

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This study is going to comprehensively examine the psychometric properties of the three depression scales (Hamilton depression scale (HAMD), Hospital anxiety and depression scale (HADS), and Beck Depression Inventory (BDI)) in stroke patients over a period of three years.

DETAILED DESCRIPTION:
This study is going to comprehensively examine the psychometric properties of the three depression scales (Hamilton depression scale (HAMD), Hospital anxiety and depression scale (HADS), and Beck Depression Inventory (BDI)) in stroke patients over a period of three years.

This study will be divided into two parts. In the first part, we will spend 3 years in recruiting 200 consecutive patients with a diagnosis of first stroke onset to compare the validity, responsiveness, and acceptability of the HAMD, HADS, and BDI. All patients will be assessed using the three depression scales and other functional measures at 14, 30, 90, 180, and 365 days after stroke.

In the second part, the inter-rater reliability of the three depression scales will be examined in the first year. Sixty chronic stroke patients will be recruited in the study.

Furthermore, the other 60 chronic stroke patients will be recruited in the second year for examining the test-retest reliability and measurement error of the three depression scales.

This study would be the first one to systematically compare the psychometric properties of the three depression scales in a long-term follow up study. The results of the study will be able to help clinicians and researchers select the most suitable depression scales for stroke patients. The results will also provide us references to develop a new depression scale, if needed, for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

patients with a diagnosis stroke ability to complete questionnaires

Exclusion Criteria:

patients with other major diseases (e.g., cancer)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2005-08; Study Completion 2008-04

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Lin Hsieh, PhD, Principal Investigator — School of Occupational Therapy, College of Medicine, National Taiwan University
Locations (1):
- School of Occupational Therapy, College of Medicine, National Taiwan University, Taipei, Taipei, Taiwan